CLINICAL TRIAL: NCT00081094
Title: Detection of Hepatocellular Carcinoma by Positron Emission Tomography With C-Acetate-11 and F-fluorodeoxyglucose-18
Brief Title: Positron Emission Tomography Using Carbon-11 Acetate and Fludeoxyglucose F 18 in Detecting Hepatocellular Carcinoma (Liver Cancer) in Patients With Known or Suspected Liver Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000358907; P30CA091842 (NIH); WU-03-0771
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; recurrent adult primary liver cancer; localized resectable adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PET scan (FDG-PET & 11C-acetate-PET) (Other): Patients will undergo routine clinical FDG-PET and research 11C-acetate-PET prior to planned surgical resection of the lesion(s) or explantation of the liver.
  Interventions: Procedure: 18F-Fluorodeoxyglucose-PET (FDG-PET); Procedure: 11Carbon-Acetate-PET

INTERVENTIONS:
Procedure: 18F-Fluorodeoxyglucose-PET (FDG-PET)
Procedure: 11Carbon-Acetate-PET

SUMMARY:
RATIONALE: Imaging procedures, such as carbon-11 acetate positron emission tomography (PET) and fludeoxyglucose F 18 PET, may improve the ability to detect hepatocellular carcinoma (liver cancer) and allow doctors to plan the most effective treatment.

PURPOSE: This clinical trial is studying how well carbon-11 acetate PET and fludeoxyglucose F 18 PET work in detecting cancer in patients with liver cancer.

ELIGIBILITY:
INCLUSION:

* Biopsy-proved HCC (stage I and II by conventional staging) or one or more of the following in a patient with clinically documented cirrhosis:
* AFP > 200 mg/dL;
* A contrast-enhancing tumor mass (>1 cm) by CT or MRI; or
* A tumor mass confirmed by arteriography.
* Patient must provide written informed consent and have completed conventional imaging and staging before initiation of PET imaging.

EXCLUSION:

* Pediatric patients under the age of 18 will be excluded from consideration from this study.
* Patients with a known prior malignancy (with the exception of basal cell carcinoma of the skin and carcinoma in situ of the cervix) within 5 years will be excluded from entry into the study. However, patients with a prior HCC thought to have a new primary or recurrent HCC are eligible.
* Pregnant and breastfeeding patients.
* Patients with poorly controlled diabetes mellitus (fasting blood glucose level > 200 mg/dL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2003-09; Primary Completion 2005-06 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Relative sensitivity and specificity of positron emission tomography (PET) scanning with carbon-11 acetate and fludeoxyglucose F 18

SECONDARY OUTCOMES:
Determine whether PET identifies additional sites of disease not detected by conventional imaging
Obtain a preliminary estimate of the impact of PET on management of patients with HCC.

CONTACTS AND LOCATIONS:
Overall Officials: William C. Chapman, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States